CLINICAL TRIAL: NCT02691715
Title: Intrauterine Saline Washing for Detection Endometrial Disease in Patients With Abnormal Uterine Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Baki Senturk, Pirincipal investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 168
Record Dates: First submitted 2016-01-28; First posted 2016-02-25 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Endometrial Disease
MeSH Terms: conditions — Uterine Diseases | interventions — Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endometrial saline plus curettage (Experimental): 5 cc saline infused to the endometrial cavity and aspirated. Then routine endometrial curettage performed for same participant.
  Interventions: Procedure: Endometrial saline plus curettage
- Endometrial curettage (Active Comparator): Only routine endometrial curettage performed
  Interventions: Procedure: Endometrial curettage

INTERVENTIONS:
Procedure: Endometrial saline plus curettage
  Arms: Endometrial saline plus curettage
Procedure: Endometrial curettage
  Arms: Endometrial curettage

SUMMARY:
Investigator will examined the diagnostic effect of the endometrial washing by saline. Because this technique more less painful and easier compared to endometrial curettage. Participants will separate into two groups. In study groups before endometrial curettage 5 cc saline infused to the endometrial cavity then aspirate and put into thin prep to examined. After this procedure routine endometrial curettage will be done. In control group only endometrial curettage will be done. Pathologic results of thin prep and curettage will compared.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal uterine bleeding

Exclusion Criteria:

* Involuntary, under 35 years old,

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Cervical cytological results according to Bethesda 2003 | 1 month
  for endometrial washing sample
Endometrial hyperplasiz classification according to World Health Organization 2013 | 1 month
  for endometrial curretage sampling

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Kamil Maternity and Pediatric Research and Training Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Moschos E, Ashfaq R, McIntire DD, Liriano B, Twickler DM. Saline-infusion sonography endometrial sampling compared with endometrial biopsy in diagnosing endometrial pathology. Obstet Gynecol. 2009 Apr;113(4):881-887. doi: 10.1097/AOG.0b013e31819b3fc7. PMID 19305334
- [Result] Rotenberg O, Renz M, Reimers L, Doulaveris G, Gebb J, Goldberg GL, Dar P. Simultaneous endometrial aspiration and sonohysterography for the evaluation of endometrial pathology in women aged 50 years and older. Obstet Gynecol. 2015 Feb;125(2):414-423. doi: 10.1097/AOG.0000000000000631. PMID 25568988
- [Result] Bese T, Demirkiran F, Guralp O, Sanioglu C, Arvas M. Transtubal transport of carcinoma cells into the peritoneal cavity after saline infusion via transcervical route in patients with endometrial carcinoma. Int J Gynecol Cancer. 2009 May;19(4):682-5. doi: 10.1111/IGC.0b013e3181a48c7f. PMID 19509571
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19305334
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Simultaneous+Endometrial+Aspiration+and+Sonohysterography+for+the+Evaluation+of+Endometrial+Pathology+in+Women+Aged+50+Years+and+Older
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Transtubal+Transport+of+Carcinoma+Cells+Into+the+Peritoneal+Cavity+After+Saline+Infusion+via+Transcervical+Route+in+Patients+With+Endometrial+Carcinoma